CLINICAL TRIAL: NCT00314535
Title: Optimization of Spectroscopic Imaging Parameters and Procedures for Prostate at 3 Tesla Using an External Probe
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EX-0002 / 22073
Record Dates: First submitted 2006-04-11; First posted 2006-04-14 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Magnetic resonance (MR) spectroscopic techniques are to be developed to obtain the best data possible at 3 Tesla (3T) for the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years of age and over

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gino Fallone, PhD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada